CLINICAL TRIAL: NCT00948610
Title: Sleep & Immune Mechanisms in Rheumatoid Arthritis: Remicade Substudy
Brief Title: Sleep and Immunity in Rheumatoid Arthritis : Remicade Substudy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michael Irwin, MD, Professor in Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NHLBI RO1 HL079955; NHLBI RO1 HL079955
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo-participant will receive placebo saline solution via IV route.
  Interventions: Drug: Remicade
- Remicade (Active Comparator): Remicade-Participant will be given 10 mg/kg of drug via IV route.
  Interventions: Drug: Remicade

INTERVENTIONS:
Drug: Remicade — Remicade/ Infliximab Study Material 10mg/kg Total Volume=250cc in saline I.V. route.
  Other Names: Infliximab

SUMMARY:
More than half of rheumatoid arthritis (RA) patients complain of sleep disturbance and this cardinal complaint is associated with fatigue, pain, and depressed mood in patient with chronic inflammatory disorder. Despite the frequency of this complaint, there is limited efforts to evaluate sleep or the abnormal increases in the expression of pro-inflammatory cytokines play a key role in the progression of RA, we hypothesize that the cytokine network is one physiological system that is associated with sleep disturbances in RA patients. Pro-inflammatory cytokines signal the central nervous system and are associated with increased symptoms of pain, fatigue, and depressed mood in rheumatic patients. The specific aims of the study are to examine the contribution of cytokines on sleep by administering a TNF antagonist vs. placebo to probe the action of pro-inflammatory cytokines on sleep in RA Patients. Examination of sleep and its consequences for pro-inflammatory cytokine activity within the framework of an observational and experimental research design will have implications for understanding the psycho-biological mechanisms that link sleep and the clinical manifestations of RA. Results from this study will guide the developments of interventions that target disordered sleep with potential effects on disability in RA.

DETAILED DESCRIPTION:
Abnormal sleep is reported by more than half of rheumatoid arthritis patients, in addition to the traditional symptoms associated with the disease, such as morning stiffness, pain, and functional debility. When recording brain activity during sleep using electroencephalography or EEG. Sleep abnormalities have been found independent of pain and thus the mechanisms to account for disordered sleep in this population are unknown. The immune system, via pro-inflammatory cytokines, plays a major role in the development of rheumatoid arthritis. Pro-inflammatory cytokines are molecules that act as signals to stimulate activity of different arms of the immune system. New medications such as remicade (infliximab) have been developed which slow disease activity by blocking the activity of these pro-inflammatory cytokines. This is done by binding to the cytokine TNF and rendering it biologically inactive. Pro-inflammatory cytokines also appear to play a role in sleep. A number of basic and human studies have found that cytokines and sleep exhibit a bi-directional relationship. However, no study to date has explored this relationship in a rheumatoid arthritis population. Thus, this research study has the potential to test whether cytokines influence sleep in rheumatoid arthritis. We will determine if a single dose of a pro-inflammatory cytokine blocking medication (remicade) affects sleep in rheumatoid arthritis patients. Interested participants will undergo an eligibility interview to review in-depth subject participation, RA diagnosis, written Consent. Following eligibility, patients will undergo a single overnight sleep assessment lasting four nights at the General Clinical Research Center. After the adaption and baseline nights, on day 3, patients will be randomized to receive either 10 mg/kg of remicade or placebo and their sleep will be subsequently monitored for two additional nights ( post-infusion 1 and post-infusion 2).

ELIGIBILITY:
Inclusion Criteria:

1. Rheumatoid arthritis patients will meet American College of Rheumatology revised criteria (Arnett, Edworthy et al. 1988). This requires at least four of the following seven criteria: 1) morning joint stiffness; 2) arthritis in 3 or more joint areas; 3) arthritis of hand joints; 4) symmetric arthritis; 5) rheumatoid nodules; 6) presence of serum rheumatoid factor and 7) changes on posteroanterior hand and wrist radiographs. In addition, criteria 1-4 must be present for at least four weeks. Subjects must be between 18 and 85 years of age.
2. If rheumatoid arthritis patients are receiving treatment with traditional disease modifying antirheumatic drugs (DMARD), such as methotrexate, sulfasalazine or hydroxychloroquine, they must be on a stable regime for one month before study and stable throughout study.
3. If rheumatoid arthritis patients have received treatment with a TNF antagonist or other biologic medication, they must be drug free for greater than 3 months.

Exclusion Criteria:

1. Steroids - Individuals currently taking greater than an equivalent of 10 mg of prednisone will be excluded given the potent anti-inflammatory effects of such medications.
2. Opioids - Individuals using multiple daily dosage schedule of opioid agents such as oxycodone (Percocet), hydrocodone (Vicodin), morphine, Dilaudid will be excluded.
3. Co-morbid medical disorders - the presence of active unstable and uncontrolled co-morbid medical conditions such as diabetes, cardiovascular diseases, and cancer will be exclusionary criteria. In particular, individuals with co-morbid inflammatory disorders such as Crohn's disease and ulcerative colitis and other autoimmune disorders will be excluded. Any uncontrolled medical condition that is deemed by the investigators to interfere with the proposed study procedures, or put the study participant at undue risk will also be considered exclusionary criteria.
4. Chronic infections - individuals with chronic infections will also be excluded because of effects on immune markers measured in study.
5. Co-morbid pain disorders - individuals with co-morbid pain disorders such as fibromyalgia will also be excluded. Individuals with fibromyalgia have been found to have sleep abnormalities as well as daytime fatigue and pain and thus could confound findings.
6. Psychiatric disorders - current conditions such as major depressive disorder, bipolar disorder and risk for suicide will also be considered exclusionary criteria.
7. Gender-based criteria - pregnant or breast-feeding women will also be excluded because of their effects on neuroendocrine systems and sleep

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Irwin, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, General Clinical Research Center, Los Angeles, California, United States

REFERENCES:
- [Background] Irwin MR, Wang M, Ribeiro D, Cho HJ, Olmstead R, Breen EC, Martinez-Maza O, Cole S. Sleep loss activates cellular inflammatory signaling. Biol Psychiatry. 2008 Sep 15;64(6):538-40. doi: 10.1016/j.biopsych.2008.05.004. Epub 2008 Jun 17. PMID 18561896
- [Background] Irwin MR, Carrillo C, Olmstead R. Sleep loss activates cellular markers of inflammation: sex differences. Brain Behav Immun. 2010 Jan;24(1):54-7. doi: 10.1016/j.bbi.2009.06.001. Epub 2009 Jun 9. PMID 19520155
- [Background] Irwin MR, Davis M, Zautra A. Behavioral Comorbidities in Rheumatoid Arthritis: A Psychoneuroimmunological Perspective. Psychiatr Times. 2008 Aug 1;25(9):1. No abstract available. PMID 19590742
- [Background] Davis MC, Zautra AJ, Younger J, Motivala SJ, Attrep J, Irwin MR. Chronic stress and regulation of cellular markers of inflammation in rheumatoid arthritis: implications for fatigue. Brain Behav Immun. 2008 Jan;22(1):24-32. doi: 10.1016/j.bbi.2007.06.013. Epub 2007 Aug 15. PMID 17706915
- See also: UCLA Cousins Center for PNI — http://www.cousinspni.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Remicade
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Remicade | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.8 (14.0) | 54.1 (13.3) | 51.5 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Slow Wave Sleep
Description: Slow wave sleep in minutes at post-infusion day 2 in placebo vs. remicade
Time Frame: Post-infusion day 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | Remicade
Number analyzed (Participants) | 10 | 10
Minutes | 82.6 (39.5) | 67.3 (38.7)

2. Secondary Outcome: Cellular Inflammation
Description: Percentage of monocytes producing interleukin-6 at post-infusion day 2 in placebo vs. remicade
Time Frame: Post-infusion day 2
Measure: Mean (Standard Deviation); unit: percentage of monocytes
Arm/Group | Placebo | Remicade
Number analyzed (Participants) | 10 | 10
percentage of monocytes | 3.6 (0.6) | 4.0 (0.6)

ADVERSE EVENTS:
Arm/Group | Placebo | Remicade
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
A number of limitations exist: the sample size was relatively small; only women were included; and the exclusive use of infliximab limits generalizability to other TNF antagonists, due to differing biochemical and mechanistic profiles.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No